CLINICAL TRIAL: NCT05114460
Title: The Ability of Vaped Marijuana to Reduce the Severity of Naloxone-Precipitated Withdrawal
Brief Title: Vaped Marijuana to Attenuate Naloxone-Precipitated Withdrawal
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The U.S. Department of Health and Human Services Office of Human Research Protections issued an FWA restriction on NYSPI research that included a pause of human subjects research as of June 23, 2023. Recruitment for this trial will not reopen.
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Jermaine D. Jones, Principal Investigator, New York State Psychiatric Institute
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 8061
Record Dates: First submitted 2021-10-05; First posted 2021-11-10 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Opioid Overdose
MeSH Terms: conditions — Opiate Overdose | interventions — Naloxone; nabiximols

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Naloxone 0 mg + MJ 0.0 mg (Placebo Comparator): Intranasal naloxone in combination with vaped marijuana
  Interventions: Drug: Naloxone; Drug: Marijuana
- Naloxone 0 mg + MJ 12.5 mg (Active Comparator): Intranasal naloxone in combination with vaped marijuana
  Interventions: Drug: Marijuana
- Naloxone 0 mg + MJ 25 mg (Active Comparator): Intranasal naloxone in combination with vaped marijuana (MJ)
  Interventions: Drug: Marijuana
- Naloxone 4 mg + MJ 0.0 mg (Active Comparator): Intranasal naloxone in combination with vaped marijuana (MJ)
  Interventions: Drug: Naloxone
- Naloxone 4 mg + MJ 12.5 mg (Experimental): Intranasal naloxone in combination with vaped marijuana (MJ)
  Interventions: Drug: Naloxone; Drug: Marijuana
- Naloxone 4 mg + MJ 25 mg (Experimental): Intranasal naloxone in combination with vaped marijuana (MJ)
  Interventions: Drug: Naloxone; Drug: Marijuana

INTERVENTIONS:
Drug: Naloxone — Intranasal Naloxone
  Arms: Naloxone 0 mg + MJ 0.0 mg; Naloxone 4 mg + MJ 0.0 mg; Naloxone 4 mg + MJ 12.5 mg; Naloxone 4 mg + MJ 25 mg
Drug: Marijuana — Vaped Marijuana
  Arms: Naloxone 0 mg + MJ 0.0 mg; Naloxone 0 mg + MJ 12.5 mg; Naloxone 0 mg + MJ 25 mg; Naloxone 4 mg + MJ 12.5 mg; Naloxone 4 mg + MJ 25 mg

SUMMARY:
The goal of the proposed, proof-of-concept study is to test the combined effects of vaporized marijuana [Delta-9-tetrahydracannabinol (THC)] with NLX as a proof of concept towards the possible development of a combined overdose reversal agent with improved tolerability.

DETAILED DESCRIPTION:
The goal of the proposed, proof-of-concept study is to test the combined effects of vaporized marijuana [Delta-9-tetrahydracannabinol (THC)] with NLX as a proof of concept towards the possible development of a combined overdose reversal agent with improved tolerability. Marijuana plant material will be obtained from the National Institutes on Drug Abuse (NIDA). In clinical studies, oral synthetic THC reduced the severity of opioid withdrawal during opioid detoxification. Clinically, cannabinoid drugs like Marinol® (oral synthetic THC), Sativex ® (nabixomols), and Cesamet® (nabilone) are used to treat nausea and vomiting, common symptoms of opioid withdrawal. This study will investigate the ability of vaporized marijuana (V-MJ) (0.00, 12.5, and 25 mg: concentration= 11.7% THC + 0.04% CBD) to reduce the severity of opioid withdrawal precipitated by intranasal (IN) NLX (0.0 and 4.0 mg). This trial will recruit healthy participants with opioid use disorder (N=16, completers). Testing will begin following stabilization on oral morphine (120 mg/day), which will continue throughout the trial. During each testing session, a single V-MJ + naloxone dose combination will be assessed (in randomized order), with 48 hours between testing sessions. Laboratory testing sessions will consist of a modified naloxone challenge procedure, which quantifies the severity of naloxone-precipitated opioid withdrawal.

ELIGIBILITY:
Inclusion Criteria:

1. 18-55 years of age.
2. Diagnostic criteria for Opioid Use Disorder (OUD) moderate-severe (304.00) as per DSM-V, including physiological dependence and not currently seeking treatment for OUD.
3. Self-reported opioid use for nontherapeutic purposes; and positive urine drug screen for opioids.
4. Physically healthy.
5. Normal body weight/Within 20% of body weight (for appropriate frame) according to 1983 Metropolitan Weight tables.
6. Able to perform study procedures.
7. Females must be either:

   1. Post-menopausal (amenorrhea for at least 12 consecutive months), surgically sterile -or
   2. Women of childbearing potential must agree to use an acceptable double-barrier method of contraception during screening and study participation.
8. Must smoke < three cannabis cigarettes three times a week (or the vaping equivalent) for the four weeks before screening.

Exclusion Criteria:

1. Seeking treatment for Opioid Use Disorder.
2. Current or history of a psychiatric condition that would affect participants' ability to provide informed consent (e.g., mood disorder with functional impairment or schizophrenia) or make participant hazardous for the participant (e.g., recent suicidal ideation) or staff (e.g., significant history of violence).
3. Current DSM-V diagnosis of substance use disorders requiring medically managed detoxification, other than OUD (e.g., alcohol or benzodiazepine dependence).
4. Medical condition resulting in chronic pain (>3 months).
5. Clinically significant abnormality on physical examination, vital signs, screening laboratory tests, or 12- lead ECG.
6. Significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, or neurologic disorder.
7. Any surgical, or medical condition that may interfere with the absorption, distribution, metabolism, or excretion of the study drugs.
8. Baseline hypotension, orthostatic hypotension or syncope, hypertension (blood pressure > 140/90), pulmonary hypertension or heart disease.
9. Any of the following values for laboratory tests:

   1. positive pregnancy test,
   2. hemoglobin < 12 g/dL in males and < 11 g/dL in females,
   3. neutrophil count < 1.0 × 109/L,
   4. platelet count < 75 × 109/L,
   5. creatinine clearance < 50 ml/min per modified Cockcroft-Gault equation,
   6. aspartate aminotransferase or alanine aminotransferase > 3.0 × upper limit of normal.
10. Hypersensitivity to opioids, history of significant adverse reactions to cannabinoids, and allergy or contraindication to any other drugs administered as a part of this investigation.
11. Use of an investigational agent within 30 days.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jermaine Jones, PhD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jones JD, Martinez S, Arout C, Haney M, Castillo F, Manubay J, Perez F, Luba RR, Comer SD. The effects of vaped cannabis on the severity of naloxone-precipitated opioid withdrawal. Exp Clin Psychopharmacol. 2025 Aug 21:10.1037/pha0000796. doi: 10.1037/pha0000796. Online ahead of print. PMID 40839512

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2 participants were enrolled however, 1 participant withdrew from the study prior to completing any of the testing sessions (i.e., periods).
Pre-assignment Details: After enrollment/admission and prior to testing participants were transition from illicit opioids onto a stable daily dose of a prescription opioid.
Groups:
- All Participants: Randomized, Within-Subjects Design
Period: Naloxone 0 mg + Marijuana 0.0 mg
Arm/Group | All Participants
Started | 1
Completed | 1
Not Completed | 0
Period: Naloxone 0 mg + Marijuana 12.5 mg
Arm/Group | All Participants
Started | 1
Completed | 1
Not Completed | 0
Period: Naloxone 0 mg + Marijuana 25 mg
Arm/Group | All Participants
Started | 1
Completed | 1
Not Completed | 0
Period: Naloxone 4 mg + Marijuana 0.0 mg
Arm/Group | All Participants
Started | 1
Completed | 1
Not Completed | 0
Period: Naloxone 4 mg + Marijuana 12.5 mg
Arm/Group | All Participants
Started | 1
Completed | 1
Not Completed | 0
Period: Naloxone 4 mg + Marijuana 25 mg
Arm/Group | All Participants
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Two participants were enrolled, however, one participant withdrew themselves from the study, prior to testing to accept a work assignment.
Groups:
- All Study Participants: Two participants were enrolled in the within-subjects trial.
Arm/Group | All Study Participants
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 39 [28 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Clinical Opiate Withdrawal Scale (COWS)
Description: Clinical Opiate Withdrawal Scale is an 11-item, clinician-administered measure designed to quantify the severity of opioid withdrawal. The COWS evaluates the severity of the following symptoms on a scale of 0-4 or 5: resting pulse rate, sweating, restlessness, pupil size, bone or joint aches, runny nose or tearing, gastrointestinal upset, tremor, yawning, anxiety, or irritability, and gooseflesh. The score on the COWS ranges from 0 to 48 points with withdrawal ratings between 5-12 considered mild, 13-24 as moderate, 25-36 as moderately severe, and >36 considered severe.
Time Frame: 4-week trial: Peak COWS score throughout the testing session for each dose combination.
Population: Data are only available from 1 participant and the other participant enrolled did not complete any testing sessions.
Measure: Number; unit: units on a scale
Arm/Group | Naloxone 0 mg + MJ 0.0 mg | Naloxone 0 mg + MJ 12.5 mg | Naloxone 0 mg + MJ 25 mg | Naloxone 4 mg + MJ 0.0 mg | Naloxone 4 mg + MJ 12.5 mg | Naloxone 4 mg + MJ 25 mg
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
units on a scale | 2 | 2 | 4 | 27 | 21 | 20

ADVERSE EVENTS:
Time Frame: All Study Participants, the 4-week Inpatient testing period.
Description: An adverse event is any unwanted experience or event occurring during the trial. An adverse event will be defined as serious whenever the outcome is fatal or life-threatening, is significantly or permanently disabling or incapacitating, requires or prolongs inpatient hospitalization, results in permanent disability, results in a congenital anomaly, or is unusual and potentially serious.
Groups:
- All Study Participants: Adverse events were assessed were collected throughout the 4-week inpatient period.
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-12-15): https://cdn.clinicaltrials.gov/large-docs/60/NCT05114460/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/60/NCT05114460/SAP_002.pdf